CLINICAL TRIAL: NCT00714402
Title: Procalcitonin Level as a Prognostic Marker and Its' Kinetics in Children With Bacterial Infections
Brief Title: Procalcitonin Level and Kinetics in Children With Bacterial Infections
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Yechiel Schlesinger, Shaare Zedek Medical Center
Other Study IDs: pct.ctil
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2009-01

CONDITIONS: Bacterial Infections; Bacteremia; Meningitis; Urinary Tract Infection; Mastoiditis; Lobar Pneumonia; Septic Arthritis; Cellulitis; Osteomyelitis
Keywords: UTI
MeSH Terms: conditions — Bacterial Infections; Bacteremia; Meningitis; Urinary Tract Infections; Mastoiditis; Pneumonia; Arthritis, Infectious; Cellulitis; Osteomyelitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — whole blood

GROUPS / COHORTS (1):
- a: children with proven of probable invasive bacterial infections

SUMMARY:
The purposes of this study are:

1. To determine whether procalcitonin level at admission of pediatric patients with bacterial infections can be used as a marker for prediction of defervescence and hospitalization length
2. To examine the kinetics of procalcitonin in pediatric patients with bacterial infections and persistent fever

ELIGIBILITY:
Inclusion Criteria:

* Positive blood, urine, synovial, bone, pleural effusion, abscess or CSF culture
* Cellulitis, lobar pneumonia, osteomyelitis,

Ages: 3 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: hospitalized patients at date of admission
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-08

PRIMARY OUTCOMES:
time to defervescence | discharge

SECONDARY OUTCOMES:
length of hospitalization | discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yechiel Schlesinger, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Pob 3235, Israel

REFERENCES:
- [Background] Le Moullec JM, Jullienne A, Chenais J, Lasmoles F, Guliana JM, Milhaud G, Moukhtar MS. The complete sequence of human preprocalcitonin. FEBS Lett. 1984 Feb 13;167(1):93-7. doi: 10.1016/0014-5793(84)80839-x. PMID 6546550
- [Background] Assicot M, Gendrel D, Carsin H, Raymond J, Guilbaud J, Bohuon C. High serum procalcitonin concentrations in patients with sepsis and infection. Lancet. 1993 Feb 27;341(8844):515-8. doi: 10.1016/0140-6736(93)90277-n. PMID 8094770
- [Background] Christ-Crain M, Stolz D, Bingisser R, Muller C, Miedinger D, Huber PR, Zimmerli W, Harbarth S, Tamm M, Muller B. Procalcitonin guidance of antibiotic therapy in community-acquired pneumonia: a randomized trial. Am J Respir Crit Care Med. 2006 Jul 1;174(1):84-93. doi: 10.1164/rccm.200512-1922OC. Epub 2006 Apr 7. PMID 16603606
- [Background] Schuetz P, Christ-Crain M, Wolbers M, Schild U, Thomann R, Falconnier C, Widmer I, Neidert S, Blum CA, Schonenberger R, Henzen C, Bregenzer T, Hoess C, Krause M, Bucher HC, Zimmerli W, Muller B; ProHOSP study group. Procalcitonin guided antibiotic therapy and hospitalization in patients with lower respiratory tract infections: a prospective, multicenter, randomized controlled trial. BMC Health Serv Res. 2007 Jul 5;7:102. doi: 10.1186/1472-6963-7-102. PMID 17615073
- [Background] Nobre V, Harbarth S, Graf JD, Rohner P, Pugin J. Use of procalcitonin to shorten antibiotic treatment duration in septic patients: a randomized trial. Am J Respir Crit Care Med. 2008 Mar 1;177(5):498-505. doi: 10.1164/rccm.200708-1238OC. Epub 2007 Dec 20. PMID 18096708
- [Background] Boussekey N, Leroy O, Alfandari S, Devos P, Georges H, Guery B. Procalcitonin kinetics in the prognosis of severe community-acquired pneumonia. Intensive Care Med. 2006 Mar;32(3):469-72. doi: 10.1007/s00134-005-0047-8. Epub 2006 Feb 14. PMID 16477418
- [Background] Seligman R, Meisner M, Lisboa TC, Hertz FT, Filippin TB, Fachel JM, Teixeira PJ. Decreases in procalcitonin and C-reactive protein are strong predictors of survival in ventilator-associated pneumonia. Crit Care. 2006;10(5):R125. doi: 10.1186/cc5036. PMID 16956405
- [Background] Hatherill M, Tibby SM, Turner C, Ratnavel N, Murdoch IA. Procalcitonin and cytokine levels: relationship to organ failure and mortality in pediatric septic shock. Crit Care Med. 2000 Jul;28(7):2591-4. doi: 10.1097/00003246-200007000-00068. PMID 10921600